CLINICAL TRIAL: NCT06414226
Title: Investigation of the Effect of Krill and Fish Oil Intake on Clinical and Biochemical Findings and Eating Behavior in Adult Individuals With Major Depression Disorders
Brief Title: Comparison of Krill and Fish Oil on Clinical and Biochemical Outcomes in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Collaborators: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Murat Açık, Associate Professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021/05-35
Record Dates: First submitted 2024-04-17; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Depression
Keywords: depression; anxiety; fish oil; krill oil; eating behavior
MeSH Terms: conditions — Depression; Anxiety Disorders; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Double-Blinded
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Krill group (Experimental): Krill oil ((n=17), (EPA=340 mg, DHA=180 mg)), The duration of the intervention was 8 weeks.
  Interventions: Dietary Supplement: Krill and Fish Oil vs. Placebo
- Fish group (Experimental): 2) fish oil ((n=17)), (EPA=360 mg, DHA=240 mg), The duration of the intervention was 8 weeks.
  Interventions: Dietary Supplement: Krill and Fish Oil vs. Placebo
- Placebo (Placebo Comparator): Placebo capsule ( (n=16), (EPA=0 mg, DHA=0 mg)). The duration of the intervention was 8 weeks.
  Interventions: Dietary Supplement: Krill and Fish Oil vs. Placebo

INTERVENTIONS:
Dietary Supplement: Krill and Fish Oil vs. Placebo — Participants were prescribed to take a daily dose of 4 capsules (4×500 mg= 2 g/day) stored at an appropriate temperature during the 8-week treatment period. The patients were informed to take 2 of the capsules in the bottle to be taken orally daily in the morning before breakfast and the other 2 capsules before dinner. The capsule bottles contained 500 mg concentrated krill oil, fish oil or placebo (empty capsule) capsules. The daily intake of EPA+DHA from krill and fish oil was determined as 520 mg and 600 mg, respectively. Krill and fish oil were obtained from Aniqnaturals Superba and Orzax Ocean company, respectively.
  Other Names: Aniqnaturals Superba Krill Oil; Ocean Fish Oil

SUMMARY:
The Omega-3 polyunsaturated fatty acids (n-3 PUFA), associated with fish oil, has been one of the most studied non-pharmacological subjects for its effect on Major Depression Disorder (MDD). However, studies comparing the effect of krill oil, on depression are limited, that has similar content and different structural forms with fish oil. This study was conducted to evaluate the effectiveness of the use of krill and fish oil on clinical effects, biochemical outcomes and eating behavior in individuals diagnosed with MDD. It was included 57 adult individuals diagnosed with MDD in the psychiatry clinic in this study. Randomization was performed after inclusion and exclusion criteria were applied in the study, and participants were included in one of three groups. These groups are; 1) krill oil ((n=17), (Eicosapentaenoic acid (EPA)=340 mg, Docosahexaenoic acid (DHA)=180 mg)), 2) fish oil ((n=17)), (EPA=360 mg, DHA=240 mg), 3) placebo ( (n=16), (EPA=0 mg, DHA=0 mg)). The duration of the intervention was 8 weeks. Anthropometric measurements, biochemical outcomes and food consumption records of the participants were taken at the beginning and end of the intervention, and Hamilton depression rating scale (HDRS), depression anxiety stress-21 (DASS-21) and food craving questionnaire (FCQ) was applied to the participants. Statistical Package for Social Sciences (SPSS) and R studio software were used for statistical analysis of the data.

DETAILED DESCRIPTION:
Introduction

Major Depressive Disorder (MDD) affects approximately 6% of the adult population worldwide each year and is the second greatest contributor to the burden of chronic disease. In the treatment of MDD, both psychotherapy and psychopharmacology are effective. However, approximately 30% of patients do not achieve definitive recovery even after several treatment attempts. Major depressive disorder can affect an individual's life as a whole and is difficult to treat due to its high rate of relapse, and it is often associated with anxiety and cardiovascular diseases (CVD), which can threaten an individual's life. It is estimated that major depression is responsible for 3% of the global burden of disease according to the World Health Organization (WHO) report and that this rate may increase to 7% by 2030. Therefore, alternatives to effective treatments and prevention strategies are urgently needed due to this increasing trend.

Omega-3 polyunsaturated fatty acids (n-3 PUFAs), identified with fish oil, became one of the most researched nutritional topics on the effects of major depressive disorder. Omega-3 polyunsaturated fatty acids are shown to be effective in cardiovascular disease (CVD) prevention due to their anti-inflammatory and cardio-protective effects. It can potentially share common mechanisms with CVD, considering factors such as increased production of pro-inflammatory cytokines, endothelial dysfunction and increases in plasma homocysteine levels, which play a role in the pathophysiology of some psychiatric disorders such as depression. It is possible that omega-3 has multiple positive effects on depression through its neurogenesis and neuroplasticity abilities, as well as having a positive effect on pathophysiological mechanisms. Appleton et al. conducted a Cochrane review to investigate the effect of n-3 PUFA supplements on depression in adults. This review included 25 studies (total 1438 participants) investigating the effect of n-3 PUFA supplements versus placebo and 1 study (40 participants) comparing n-3 PUFA supplements with antidepressant treatment. As a result, it was reported that n-3 PUFA supplements had a modestly positive effect on depression compared to placebo. However, it was emphasized in this report that the majority of the studies (22 studies) had a low level of evidence. This was attributed to factors such as high levels of bias, duration of follow-up, methodological errors and deficiencies due to blinded designs. The general conclusion of the authors was that there was a need for high quality intervention studies in this field.

Although there are a large number of studies focusing on the use of fish oil in depression, research using krill oil, another source rich in n-3 PUFAs, is very limited. Krill oil is an important shellfish that lives in the oceans around the Antarctic continent and attracts attention in research due to its rich omega-3 fatty acid content. As krill is a species living in cold regions, they are rich in EPA and DHA content, along with PUFAs in the form of phospholipids and especially phosphatidylcholine in cell membrane structures. The form containing and binding Docosahexaenoic acid (DHA) and Eicosapentaenoic acid (EPA) in krill oil is phospholipids, contrary to triglyceride in fish oil. Therefore, the absorption and bioavailability activities are different because of the difference in the forms in fish and krill oil. Although there are studies on the effects of krill oil on the nervous system on the human research, there is limited research on the effectiveness of krill oil on depression. To our knowledge, there was only one pilot study on rats comparing the treatment efficacy of fish and krill oil on depression. This study compared the antidepressant effects of krill (EPA: 60 mg/500 mg, DHA: 35 mg/500 mg) and fish oil (EPA: 90 mg/500 mg, DHA: 60 mg/500 mg), vitamin B12 and imipramine. As a result, krill oil showed favorable results on a number of variables compared to fish oil, but similar results were found in both groups. It is important to compare the efficacy of krill and fish oil with similar EPA and DHA content on depression to clarify the question of which of these oils in different forms may be more effective on the disease.

Major depressive disorders affect many mechanisms such as food intake, taste perception and food selection. When clinical pictures related to the nutritional status of depressed individuals are examined; changes in appetite, increased consumption of certain food groups and related changes in body weight are frequently observed. In addition, antidepressant drugs used may also affect food intake and weight control. Eating behavior is under the control of complex neural mechanisms, especially serotonin. At the same time, food intake is also effective in the control of serotonin release in serotonergic neurons. Serotonin, which has a bidirectional relationship with eating behavior, is a neurotransmitter involved in the physiopathology of many psychiatric disorders. The presence of a disorder in the serotonin pathway may explain the development of both psychiatric disorders and obesity in the patient. As a result, it was reported that eating behavior disorders, interest in unhealthy food consumption and increased appetite in major depressives, as in some psychiatric disorders, may lead to an increase in body weight in individuals during the illness or in progressive processes. There are several studies examining the relationship between depression and obesity. However, clinical studies to determine the factors leading to this condition are limited. In addition, data collection on eating behavior, appetite and weight status is neglected in most clinical interventions in patients with depression. Therefore, it is important to investigate the efficacy of n-3 fatty acids on appetite and body composition as well as eating behaviors that examine food cravings in depressed individuals.

Considering all of these opinions, this study aimed to determine the effectiveness of krill and fish oil on clinical effects, biochemical findings and eating behavior in individuals diagnosed with MDD and to compare the results with the control group.

METHODS

This study was designed with a randomized double-blind placebo-controlled. The study was conducted in the Psychiatry Clinic of Adıyaman University Training and Research Hospital with 50 patients over the age of 18 diagnosed with MDD. The duration of the intervention for each participant was 8 weeks. The included patients received fish oil or krill oil or placebo. The study was conducted in accordance with good clinical guidelines and in accordance with the Declaration of Helsinki. Ethical approval was also obtained from the Ethics Committee of Fırat University.

Participants

The study was enrolled with 66 patients with MDD who were over 18 years of age and fulfilled the inclusion criteria. Inclusion criteria were; 1) being diagnosed with major depression by a psychiatrist in accordance with DSM V diagnostic criteria 2) not taking antidepressant medication or being on antidepressant medication for the last 1 month without medication change 3) signing the informed consent form. The exclusion criteria were as follows; 1) those who used more than two antidepressants 2) substance users in the last 6 months 3) alcohol dependence 4) suicidal ideation and suicidal tendencies (followed up by clinicians) 5) presence of other psychiatric disorders such as comorbid psychosis, schizophrenia and bipolar (excluding dysthymia and anxiety) 6) Presence of serious chronic diseases 7) pregnant or lactating women 8) Medication users that may cause emotional symptoms (Escitoloprom/Lexopro etc.) 9) food allergies 10) individuals at high risk of bleeding or those taking anti-coagulant drugs such as warfarin 11) Consumers of 3 or more servings of fish per week 12) Using any nutritional supplement 13) Hypercholesterolemia or taking medication for hypercholesterolemia 14) those who did not sign the informed consent form.

Sample Size and Randomization and Blinded

The sample size was determined based on the findings of a similar study, using the G* power 3.1.9.7 software program with an effect size of 0.224, 95% confidence interval, and a margin of error of 0.05.

This study was a randomized controlled double-blind study design. The assignment of patients to groups (randomization) was performed by a statistician who was not involved in the research and was concealed from the patients. At the first stage, stratified randomization was performed to ensure homogeneous distribution of patients according to age and gender, and then simple randomization was performed from each layer to ensure equal assignment to all groups. Each patient was assigned a number between 1-60 and then stratified according to gender (male and female) and age group (18-34 and 35-64 years). In the last stage, numbers were generated with the R studio statistical program to assign an equal number of patients to each group.

The statistician randomly assigned the color codes on the capsule bottles to each group and each group received the test products from the researcher in a closed package according to the color codes. These color codes were not known by the researchers and patients until the endpoint of the study. In addition, the researcher, clinician, and participant were blinded until the study was reported.

Intervention

The researcher conducted three 45-minute interviews with the participants for 8 weeks at the beginning, mid and end of the study. In the first interview, patients were given the product they should receive for 8 weeks in closed boxes.

Hamilton Depression Rating Scale in the questionnaire form was completed by the clinician to assess the degree of depression and clinical status of the participants. Then, the remaining parts of the questionnaire were directed to the patients. Anthropometric measurements were performed after completion of the questionnaire. Blood samples were collected from participants at the beginning and end of the study to analyze biochemical outcomes. The second interview was conducted at mid-study at the end of week 4 and the final interview was conducted at the end of week 8. In the second interview with the patients, the same procedures were performed except for the collection of blood samples and the food craving scale. In the last interview, the protocols were the same except for product administration.

Participants were prescribed a daily dose of 4 capsules (4×500 mg= 2 g/day) stored at the appropriate temperature during the 8-week treatment period. Patients were informed to take 2 of the capsules in the daily oral bottle in the morning before breakfast and the other 2 capsules before dinner. The capsule bottles contained 500 mg concentrated krill oil, fish oil or placebo capsules. The daily intake of EPA+DHA from krill and fish oil was determined as 520 mg and 600 mg, respectively.

Data Collection

Data of the participants were collected at the beginning, middle and end of the study, three times in total, by face-to-face interview with a questionnaire form. The questionnaire included sociodemographic characteristics, health information, lifestyle, Hamilton Depression Rating Scale, Depression-Anxiety-Stress Scale, Food Cravings Scale, anthropometric measurements and one-day food consumption record.

Statistical Analysis

Statistical Package for Social Sciences (SPSS) and R studio software program were used for statistical analysis of the data. The mean and standard deviation values were given for continuous data that met the normal distribution condition, otherwise the median and quartiles (25th and 75th quartile values) were given. Categorical data were presented as frequency and percentage. One-way ANOVA test was used to compare continuous variables that met the normal distribution condition between the groups, and Kruskal-Wallis H test was used for those that did not meet the normal distribution condition. Pearson chi-square test was used to compare categorical data. Repeated measures ANOVA (General linear model) test was used in the comparison of more than two dependent variables if they met the normal distribution condition. To evaluate the differences between groups, p time, p group and p group×time interaction effect were shown. The p time value expresses the comparison of any numerical variable in the group between times. The p time×groups value expresses the comparison of the numerical variable between the groups depending on time. In other words, it gives information about whether the study groups have superiority over each other during the intervention period on any variable. In addition, partial eta square values are presented for the effect size of the interaction effect of group and time. A partial eta squared value of <0.06 indicates a "small" effect size, a value between 0.06-0.14 indicates a "medium" effect size and a value >0.14 indicates a "large" effect size. In addition, the standardized mean differences, standard error, 95% confidence interval and p-values of the participants' depression, anxiety and stress scores within each group were presented. Bonferroni correction was used to calculate the p-value. If the normal distribution condition was not met, Friedman test was used and if p<0.05, Wilcoxon test was performed in paired groups and Bonferroni correction was used to calculate the p value. In addition, after the classification of depression, anxiety and stress within the groups, the Stuart-Maxwell test (R studio) was used to test the statistical significance of the changes in the severity of the disease before and after the intervention. The results were evaluated at 95% confidence intervals and a pairwise p<0.05 was considered statistically significant.

References

1. Bromet, E., et al., Cross-national epidemiology of DSM-IV major depressive episode. BMC medicine, 2011. 9: p. 1-16.
2. Rush, A.J., et al., Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR* D report. Focus, 2008. 6(1): p. 128-142.
3. Thase, M.E., et al., Cognitive Therapy Versus Medication in Augmentation and Switch Strategies as Second-Step Treatments: A STAR* D Report. Focus, 2008. 6(1): p. 104-119.
4. Organization, W.H., Depression. Fact sheet No. 369/October 2012. 2015.
5. Rangel-Huerta, O.D. and A. Gil, Omega 3 fatty acids in cardiovascular disease risk factors: An updated systematic review of randomised clinical trials. Clinical nutrition, 2018. 37(1): p. 72-77.
6. Buoite Stella, A., et al., Update on the impact of omega 3 fatty acids on inflammation, insulin resistance and sarcopenia: a review. International journal of molecular sciences, 2018. 19(1): p. 218.
7. Crupi, R., A. Marino, and S. Cuzzocrea, n-3 fatty acids: role in neurogenesis and neuroplasticity. Current medicinal chemistry, 2013. 20(24): p. 2953-2963.
8. Appleton, K.M., et al., Omega-3 fatty acids for depression in adults. Cochrane Database of Systematic Reviews, 2021(11).
9. Burri, L., Krill oil supplementation and cognitive function, in Diet and Nutrition in Dementia and Cognitive Decline. 2015, Elsevier. p. 1031-1038.
10. Colletti, A., et al., Advances in technologies for highly active omega-3 fatty acids from krill oil: Clinical applications. Marine Drugs, 2021. 19(6): p. 306.
11. Adıgüzel, K.T., K. Işgın, and G. Pekcan, Krill yağı desteği ve yeni bilimsel kanıtlar. Beslenme ve Diyet Dergisi, 2015. 43(3): p. 258-263.
12. Di Marzo, V., et al., Dietary krill oil increases docosahexaenoic acid and reduces 2-arachidonoylglycerol but not N-acylethanolamine levels in the brain of obese Zucker rats. International dairy journal, 2010. 20(4): p. 231-235.
13. Konagai, C., et al., Effects of krill oil containing n-3 polyunsaturated fatty acids in phospholipid form on human brain function: a randomized controlled trial in healthy elderly volunteers. Clinical interventions in aging, 2013: p. 1247-1257.
14. Zadeh-Ardabili, P.M., et al., Antidepressant-like effects of fish, krill oils and Vit B12 against exposure to stress environment in mice models: current status and pilot study. Scientific reports, 2019. 9(1): p. 19953.
15. Wurtman, R.J. and J.J. Wurtman, Brain serotonin, carbohydrate-craving, obesity and depression. Obesity research, 1995. 3(S4): p. 477S-480S.
16. Paans, N.P., et al., Depression and eating styles are independently associated with dietary intake. Appetite, 2019. 134: p. 103-110.
17. Lopresti, A.L., S.D. Hood, and P.D. Drummond, A review of lifestyle factors that contribute to important pathways associated with major depression: diet, sleep and exercise. Journal of affective disorders, 2013. 148(1): p. 12-27.
18. SM, S., Stahl'ın temel psikofarmakolojisi: nörobilimsel ve pratik uygulamalar. Cambridge University Press. T Uzbay (çev. ed.), 2012. 3: p. 535-6.
19. Blaine, B., Does depression cause obesity? A meta-analysis of longitudinal studies of depression and weight control. Journal of health psychology, 2008. 13(8): p. 1190-1197.
20. Luppino, F.S., et al., Overweight, obesity, and depression: a systematic review and meta-analysis of longitudinal studies. Archives of general psychiatry, 2010. 67(3): p. 220-229.
21. Lespérance, F., et al., The efficacy of omega-3 supplementation for major depression: a randomized controlled trial. Journal of Clinical Psychiatry, 2011. 72(8): p. 1054.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 19-65 years
* To be diagnosed with major depression by a psychiatrist in accordance with DSM V diagnostic criteria
* Not taking antidepressant medication or being on antidepressant medication for the last 1 month without medication change
* To have signed the informed voluntary consent form.

Exclusion Criteria:

* More than two antidepressants
* Substance users in the last 6 months
* Those with alcohol addiction
* Suicidal ideation and suicidal behaviour (followed up by clinicians)
* Presence of other psychiatric disorders such as psychosis, schizophrenia and bipolar (except dysthymia and anxiety)
* Presence of serious chronic diseases
* Women during pregnancy or lactation
* People taking medication that may cause emotional symptoms (Escitoloprom/Lexopro etc.)
* Food allergy
* Individuals at high risk of bleeding or taking anti-coagulant medication such as warfarin
* Consuming 3 portions of fish or more per week
* Use of any nutritional supplements
* People with hypercholesterolaemia or taking medication for hypercholesterolaemia

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Results of Clinical Findings | At baseline, At the end of 4th week and At the end of 8th week
  Hamilton Depression Rating Scale (HDRS): The HDRS focuses more on melancholic and physical symptoms of depression. In the HDRS, which consists of twenty-one questions, a score is calculated by answering 17 questions. The items of the scale related to difficulty falling asleep, waking up in the middle of the night, waking up early in the morning, somatic symptoms, genital symptoms, weakening and insight are graded between "0-2" and the other items are graded between "0-4". In the scale; 0-7 points: "no depression", 8-17 points: "mild depression", 18-24 points: "moderate depression" and >23 points: "severe depression".
Results of Clinical Findings | At baseline, At the end of 4th week and At the end of 8th week
  Depression Anxiety Stress Scale-21 (DASS-21): Depression Anxiety Stress Scale-21 consists of a total of 21 items aiming to measure depression, anxiety and stress levels. An individual's score of 5 points or more from the depression sub-dimension, 4 points or more from anxiety, and 8 points or more from stress indicates that he/she has the related problem.

SECONDARY OUTCOMES:
Biochemical Outcomes | At baseline and At the end of 8th week
  Biochemical Outcome: Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) Alkaline phosphatase (ALP), Gamma-glutamyltransferase (GGT), Glucose, HbA1c, Blood urea nitrogen (BUN), Creatine, Uric acid, Total cholesterol (Total-c), Triglycerides, Low density lipoprotein (LDL)-c, High density lipoprotein (HDL-c), Sodium (Na), Potassium (K), Calcium (Ca), Iron (Fe), Iron binding capacity (IBC)
Height | At baseline, At the end of 4th week and At the end of 8th week
  Anthropometric Measurements: Height (cm) will be measured with a non-flexible tape measure while standing in the frankfort plane (feet side by side with the heel and occipital region touching the wall). The body fat percentage (%), body lean mass (kg) and body fluid (%) of the individuals will be determined via a body analyzer.
Dietary Intake | At baseline and At the end of 8th week
  24-hour dietary record
Body weight | At baseline, At the end of 4th week and At the end of 8th week
  In the study, body weight (kg) measurements of the individuals participating will be measured by the researcher.
BMI | At baseline, At the end of 4th week and At the end of 8th week
  Body mass index (kg/m2) will be calculated by dividing the square of height by body weight.

OTHER OUTCOMES:
Evaluation of Eating Behaviour of the Study | At baseline and At the end of 8th week
  Food Cravings Questionnaire Scale: The FCQ scale consists of 39 items and 9 factors.Sub-dimensions of the scale; intention and planning to consume food (3 items), expectation of positive reinforcement that may arise from eating, expectation of relief from negative situations and emotions arising from eating, the possibility of lack of eating control if food is eaten, preoccupation with food and thoughts, craving as a physiological domain, feelings that may be experienced before or during the desire to eat or eating, cues that may trigger the desire to eat, guilt that may be experienced as a result of giving in to desire and/or craving. All of the items in the scale are 6-point Likert type. The score of the scale is obtained by dividing the total item scores by the number of items. The scores obtained in this way express the high desire to eat in the overall scale and sub-dimensions (Cepeda-Benito et al., 2000 and Müftüoğlu, 2016).

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University Training and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided